CLINICAL TRIAL: NCT01230281
Title: A Study to Evaluate Pharmacokinetics of C3G and to Estimate Antioxidative Markers After Repeated Administration of Black Bean Seed Coat Extract
Acronym: C3G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Rural Development Administration, Korea (Unknown)
Responsible Party: Dong-Seok Yim, Seoul St. Mary's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CPT2010-06
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-10

CONDITIONS: Oxidative Stress
Keywords: C3G; Oxidative stress; Antioxidant; Black bean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Black bean seed coat extract (Experimental): Daily 1000 mg oral Black bean seed coat extract is given to each subject for 2 weeks from Day2 after measuring antioxidative marker without intervention on Day1.
  Interventions: Other: Black bean seed coat extract

INTERVENTIONS:
Other: Black bean seed coat extract — 1000 mg oral daily dose for 2 weeks

SUMMARY:
This study is to evaluate pharmacokinetic-pharmacodynamic property of C3G after administration of Mulberry fruit extract to 12 healthy Korean volunteers. Plasma concentration of C3G and the antioxidative markers such as total antioxidative capacity and attack of free oxygen radical will be measured.

Additional objective is to investigate the multiple dose (2 weeks) safety of daily 1000mg black bean seed coat extract.

This study, as an exploratory trial, does not required statistical hypothesis

ELIGIBILITY:
Inclusion Criteria:

* Body weight >55 kg for male, >45 kg for female (within 80-120% of Ideal body weight)
* Give written informed consent and voluntarily decide participation

Exclusion Criteria:

* Acute or chronic disease symptom on screening
* Existing active and clinically significant disease involving more than one organ system
* Known allergy to Mulberry or other berries
* Positive drug or alcohol screening
* Smokers of 10 or more cigarettes per day
* Participation in a clinical trial during last 2 month prior to the start of the study
* Pregnancy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cmax - Maximum Observed Concentration - C3G in Plasma | Blood samples collected over 6 hours
AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated) - C3G in Plasma | Blood samples collected over 6 hours
Antioxidative markers | 2 weeks

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Seok Yim, M.D., PhD., Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St.Mary's Hospital, Seoul, South Korea